CLINICAL TRIAL: NCT07214506
Title: Human Papillomavirus Self-Sampling Options to Promote Equity (HOPE)
Brief Title: Human Papillomavirus (HPV) Self-Sampling Options to Promote Equity
Acronym: HOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH); El Rio Santa Cruz Neighborhood Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00007058; 5P30CA023074-43 (NIH)
Record Dates: First submitted 2025-10-07; First posted 2025-10-09 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Uterine Cervical Neoplasms; HPV Testing; Pap Smear
Keywords: Cervical cancer screening; HPV self-collection; HPV test; Mobile health unit; Unhoused individuals; Community outreach
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Papanicolaou Test

STUDY DESIGN:
Intervention Model Description: The proposed trial will randomize eight of the street medicine team's outreach sites 1:1 to either the intervention (invitation to Human Papillomavirus self-collection for cervical cancer screening in the mobile health unit plus usual care from the street medicine team) or usual care alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Human papillomavirus self-collection for Cervical Cancer Screening (Experimental): The eight outreach sites will be randomized 1:1 to arm 1 (invitation to human papillomavirus self-collection in the mobile health unit) or arm 2 (usual care), stratifying on type of outreach site to ensure balance between shelter and encampment sites in both arms.
  Interventions: Other: Human papillomavirus Self-collection
- Usual Care (Active Comparator): The eight outreach sites will be randomized 1:1 to arm 1 (invitation to HPV self-collection in the MHU) or arm 2 (usual care), stratifying on type of outreach site to ensure balance between shelter and encampment sites in both arms
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Human papillomavirus Self-collection — The individual will receive both verbal instruction on self-collection from trained health educators in the mobile health unit, as well as adapted educational materials on human papillomavirus self-collection and information about follow-up care in the case of abnormal results. Individuals will be provided with a safe and private space in the Mobile Health Unit to self-collect.
  Other Names: HPV self-sampling
  Arms: Human papillomavirus self-collection for Cervical Cancer Screening
Other: Usual Care — Usual care, will involve reminders about overdue Cervical Cancer screening and support with scheduling clinic appointments for screening, arranging for transportation, and addressing other barriers to attendance
  Other Names: Pap smear; HPV/PAP Co-test; Provider Sampling
  Arms: Usual Care

SUMMARY:
This study is testing a new way to help people who are unhoused get screened for cervical cancer. Cervical cancer can often be prevented if it is found early. Many people who lack stable housing usually do not receive regular screenings.

Through this project, the investigators will bring screening to community locations in Tucson, Arizona, using a mobile health unit (MHU) from the University of Arizona (UA) and El Rio Health. At these sites, participants will receive easy-to-understand education about cervical cancer, learn how to collect their own sample for human papillomavirus (HPV) testing, and get follow-up care if needed.

The study has two goals:

* First, the investigators will see if this community-based approach helps more people complete cervical cancer screening.
* Second, the investigators will ask participants, clinicians, and outreach staff for their opinions about the program and its practicality and acceptability.

By testing this approach, the investigators hope to find a way to make cervical cancer screening more accessible and effective for unhoused individuals.

DETAILED DESCRIPTION:
Cervical cancer can often be prevented if it is found early, but many unhoused people don't get regular screening. Through this project, the investigators are offering cervical cancer screening in community settings, such as our mobile health units, to make access easier.

Our proposal aims to design and pilot test an human papillomavirus (HPV) self-sampling program run through an MHU (operated by the UA) throughout El Rio's established outreach sites to people who are unhoused and residing in shelters and outdoor encampments. The proposed intervention, delivered through a clinic-community linkage, will include tailored education about the importance of cervical cancer screening, information on how to perform HPV self-collection, and follow-up as needed. The investigators propose the following Aims:

Aim 1. In a pragmatic pilot trial, assess the preliminary effectiveness of a community-driven, resource-efficient MHU-delivered program to distribute HPV DNA self-collection test kits to eligible unhoused individuals in Tucson, Arizona.

The primary outcome will be the completion of screening among eligible individuals. Secondary outcomes will be (1) screening modality selected (self-collected HPV, clinician-collected HPV, Pap smear, or co-test) and (2) follow-up of abnormal initial screening results within 6 months after the initial result.

Aim 2. Evaluate the feasibility and acceptability of the MHU-based HPV self-collection program through in-depth interviews with individuals who completed self-collection, clinicians, and outreach staff in the HOPE program.

Interview domains will be informed by the COM-B (capability, opportunities, motivation - behavior) framework, and outcomes will be analyzed using thematic analysis with a combination of inductive and deductive coding.

ELIGIBILITY:
Inclusion Criteria:

* Women or transgender men with a cervix
* Ages 30-64 years
* Due for cervical cancer screening:

  1. No Pap test in the past 3 years, or
  2. No human papillomavirus (HPV) test in the past 5 years
* Unhoused or unstably housed

Exclusion Criteria:

* History of cervical cancer
* HIV positive
* History of total hysterectomy
* Known pregnancy

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cervical Cancer Screening Completion | From enrollment to the end of treatment at 8 weeks
  Cervical cancer screening completion will be defined as the completion of any form of cervical cancer screening permitted according to the U.S. Preventive Services Task Force (USPSTF) guidelines, including Pap tests, Pap tests with high-risk human papillomavirus tests (cotesting), or high-risk human papillomavirus testing alone. The primary outcome will be assessed within 2 months of the street medicine team's patient contact during the trial period to account for the time required for scheduling a clinic appointment.

SECONDARY OUTCOMES:
Follow-up adherence | From identification of abnormal results to 6 months
  The secondary outcome will be follow-up adherence for abnormal screening results ascertained via electronic health record review within six months of the abnormal result

CONTACTS AND LOCATIONS:
Overall Officials: Dan Theodorescu, MD, PhD, Principal Investigator — University of Arizona; Purnima Madhivanan, MBBS, MPH, PhD, Study Chair — University of Arizona
Locations (1):
- El Rio Santa Cruz Neighborhood Health, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
HOPE Project Resource and Data Sharing Plan Resource and data sharing are central to the goals of the National Institutes of Health (NIH) and support open science, collaboration, and the translation of research results into improved public health. The HOPE project (HPV Self-Sampling Options to Promote Equity) will follow NIH policies for responsible data sharing, ensuring participant confidentiality and adherence to all Health Insurance Portability and Accountability Act (HIPAA) rules.
  Commitment to Dissemination The HOPE project team is committed to the timely and open dissemination of study findings. Results will be shared with community partners, policymakers, and the scientific community through peer-reviewed journal publications, conference presentations, newsletters, and community forums. All publications will adhere to the NIH Public Access Policy guidelines, with manuscripts submitted to PubMed Central. Findings will also be presented at relevant national and international con
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months after publication, with no end date
Access Criteria: Any researcher seeking access to HOPE data who submits a written request describing the purpose, planned analyses, and data security measures

REFERENCES:
- [Background] Brown AW, Li P, Bohan Brown MM, Kaiser KA, Keith SW, Oakes JM, Allison DB. Best (but oft-forgotten) practices: designing, analyzing, and reporting cluster randomized controlled trials. Am J Clin Nutr. 2015 Aug;102(2):241-8. doi: 10.3945/ajcn.114.105072. Epub 2015 May 27. PMID 26016864
- [Background] Li P, Redden DT. Small sample performance of bias-corrected sandwich estimators for cluster-randomized trials with binary outcomes. Stat Med. 2015 Jan 30;34(2):281-96. doi: 10.1002/sim.6344. Epub 2014 Oct 24. PMID 25345738
- [Background] Heintzman J, Hatch B, Coronado G, Ezekiel D, Cowburn S, Escamilla-Sanchez O, Marino M. Role of Race/Ethnicity, Language, and Insurance in Use of Cervical Cancer Prevention Services Among Low-Income Hispanic Women, 2009-2013. Prev Chronic Dis. 2018 Feb 22;15:E25. doi: 10.5888/pcd15.170267. PMID 29470167
- [Background] US Preventive Services Task Force; Curry SJ, Krist AH, Owens DK, Barry MJ, Caughey AB, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Kubik M, Landefeld CS, Mangione CM, Phipps MG, Silverstein M, Simon MA, Tseng CW, Wong JB. Screening for Cervical Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2018 Aug 21;320(7):674-686. doi: 10.1001/jama.2018.10897. PMID 30140884
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Sabatino SA, Thompson TD, White MC, Shapiro JA, Clarke TC, Croswell JM, Richardson LC. Cancer Screening Test Use-U.S., 2019. Am J Prev Med. 2022 Sep;63(3):431-439. doi: 10.1016/j.amepre.2022.02.018. Epub 2022 Apr 22. PMID 35469700
- [Background] Christian NJ, Havlik J, Tsai J. The Use of Mobile Medical Units for Populations Experiencing Homelessness in the United States: A Scoping Review. J Gen Intern Med. 2024 Jun;39(8):1474-1487. doi: 10.1007/s11606-024-08731-9. Epub 2024 Mar 25. PMID 38528232
- [Background] Degife EA, Oliveira CR, Znamierowski E, Meyer JP, Sheth SS. Uptake of Cervical Cancer Screening Among Female Patients Using a Mobile Medical Clinic. Am J Prev Med. 2023 Nov;65(5):835-843. doi: 10.1016/j.amepre.2023.05.013. Epub 2023 May 21. PMID 37220860
- [Background] Greenwald ZR, El-Zein M, Bouten S, Ensha H, Vazquez FL, Franco EL. Mobile Screening Units for the Early Detection of Cancer: A Systematic Review. Cancer Epidemiol Biomarkers Prev. 2017 Dec;26(12):1679-1694. doi: 10.1158/1055-9965.EPI-17-0454. Epub 2017 Oct 4. PMID 28978564
- [Background] De Mil R, Guillaume E, Launay L, Guittet L, Dejardin O, Bouvier V, Notari A, Launoy G, Berchi C. Cost-Effectiveness Analysis of a Mobile Mammography Unit for Breast Cancer Screening to Reduce Geographic and Social Health Inequalities. Value Health. 2019 Oct;22(10):1111-1118. doi: 10.1016/j.jval.2019.06.001. Epub 2019 Jul 29. PMID 31563253
- [Background] Pretsch PK, Spees LP, Brewer NT, Hudgens MG, Sanusi B, Rohner E, Miller E, Jackson SL, Barclay L, Carter A, Wheeler SB, Smith JS. Effect of HPV self-collection kits on cervical cancer screening uptake among under-screened women from low-income US backgrounds (MBMT-3): a phase 3, open-label, randomised controlled trial. Lancet Public Health. 2023 Jun;8(6):e411-e421. doi: 10.1016/S2468-2667(23)00076-2. Epub 2023 May 11. PMID 37182529
- [Background] Winer RL, Lin J, Anderson ML, Tiro JA, Green BB, Gao H, Meenan RT, Hansen K, Sparks A, Buist DSM. Strategies to Increase Cervical Cancer Screening With Mailed Human Papillomavirus Self-Sampling Kits: A Randomized Clinical Trial. JAMA. 2023 Nov 28;330(20):1971-1981. doi: 10.1001/jama.2023.21471. PMID 38015219
- [Background] Winer RL, Lin J, Tiro JA, Miglioretti DL, Beatty T, Gao H, Kimbel K, Thayer C, Buist DSM. Effect of Mailed Human Papillomavirus Test Kits vs Usual Care Reminders on Cervical Cancer Screening Uptake, Precancer Detection, and Treatment: A Randomized Clinical Trial. JAMA Netw Open. 2019 Nov 1;2(11):e1914729. doi: 10.1001/jamanetworkopen.2019.14729. PMID 31693128
- [Background] Bharel M, Casey C, Wittenberg E. Disparities in cancer screening: acceptance of Pap smears among homeless women. J Womens Health (Larchmt). 2009 Dec;18(12):2011-6. doi: 10.1089/jwh.2008.1111. PMID 20044864
- [Background] Asgary R. Cancer screening in the homeless population. Lancet Oncol. 2018 Jul;19(7):e344-e350. doi: 10.1016/S1470-2045(18)30200-6. Epub 2018 Jun 29. PMID 30084381
- [Background] Chau S, Chin M, Chang J, Luecha A, Cheng E, Schlesinger J, Rao V, Huang D, Maxwell AE, Usatine R, Bastani R, Gelberg L. Cancer risk behaviors and screening rates among homeless adults in Los Angeles County. Cancer Epidemiol Biomarkers Prev. 2002 May;11(5):431-8. PMID 12010856
- [Background] Long HL, Tulsky JP, Chambers DB, Alpers LS, Robertson MJ, Moss AR, Chesney MA. Cancer screening in homeless women: attitudes and behaviors. J Health Care Poor Underserved. 1998 Aug;9(3):276-92. doi: 10.1353/hpu.2010.0070. PMID 10073209
- [Background] Huntington S, Puri Sudhir K, Schneider V, Sargent A, Turner K, Crosbie EJ, Adams EJ. Two self-sampling strategies for HPV primary cervical cancer screening compared with clinician-collected sampling: an economic evaluation. BMJ Open. 2023 Jun 6;13(6):e068940. doi: 10.1136/bmjopen-2022-068940. PMID 37280031
- [Background] Kohler RE, Roncarati JS, Aguiar A, Chatterjee P, Gaeta J, Viswanath K, Henry C. Trauma and cervical cancer screening among women experiencing homelessness: A call for trauma-informed care. Womens Health (Lond). 2021 Jan-Dec;17:17455065211029238. doi: 10.1177/17455065211029238. PMID 34225506
- [Background] Jeleff M, Haider S, Schiffler T, Gil-Salmeron A, Yang L, Barreto Schuch F, Grabovac I. Cancer risk factors and access to cancer prevention services for people experiencing homelessness. Lancet Public Health. 2024 Feb;9(2):e128-e146. doi: 10.1016/S2468-2667(23)00298-0. PMID 38307679
- [Background] The 2023 Annual Homelessness Assessment Report. US Department of Housing and Urban Development. Published online December 2023. Accessed December 6, 2024. https://www.huduser.gov/portal/sites/default/files/pdf/2023-AHAR-Part-1.pdf
- [Background] Baggett TP, Chang Y, Porneala BC, Bharel M, Singer DE, Rigotti NA. Disparities in Cancer Incidence, Stage, and Mortality at Boston Health Care for the Homeless Program. Am J Prev Med. 2015 Nov;49(5):694-702. doi: 10.1016/j.amepre.2015.03.038. Epub 2015 Jul 3. PMID 26143955